CLINICAL TRIAL: NCT03125863
Title: Acute Hemostasis Following the Use of the AQUABEAM® System for the Treatment of Benign Prostatic Hyperplasia
Acronym: AHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0113
Record Dates: First submitted 2016-08-09; First posted 2017-04-24 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Image-guided; BPH; Aquablation; AQUABEAM; LUTS; Tissue resection; Robotics
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive treatment with the AquaBeam System to remove enlarged prostatic tissue. Following the aquablation intervention, a urinary catheter will be inserted to apply pressure on treated tissue for hemostasis.
  Interventions: Device: AquaBeam System

INTERVENTIONS:
Device: AquaBeam System — The AquaBeam system delivers a high-velocity saline stream under precise electromechanical control and live ultrasound guidance to ablate prostatic glandular tissue without the production of heat. The physician uses ultrasound imaging to plan the treatment contour and depth to define the treatment region. The AquaBeam ablates the target tissue, adhering to the pre-defined treatment zone.

SUMMARY:
A single-arm prospective, interventional clinical trial to evaluate the safety and performance of obtaining hemostasis with commercially approved catheters following prostate resection using the AquaBeam for treatment of LUTS resulting from BPH.

DETAILED DESCRIPTION:
PROCEPT BioRobotics has developed the AquaBeam, a personalized image-guided waterjet resection system that utilizes a high-velocity saline stream to resect and remove prostate tissue in males suffering from Lower Urinary Tract Symptoms (LUTS) due to BPH. The AquaBeam System is intended for the resection and removal of prostate tissue in patients experiencing LUTS. The primary objective of the study is to evaluate the safety and performance of obtaining hemostasis with commercially approved catheters following prostate resection using the AquaBeam. The time frame of the study is 7 days. Up to 30 participants will be included in this single-site clinical trial. The trial is a single-arm prospective, interventional clinical study. Results will be analyzed to determine the safety and efficacy of commercially approved catheters for the achievement of acute hemostasis without the need for cauterization.

ELIGIBILITY:
Inclusion Criteria:

* Male age from 40 through 85 years with LUTS due to BPH

Exclusion Criteria:

* Any severe illness that would prevent complete study participation or confound study results

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2016-09-03 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Completion of the intended surgical procedure | 7 days post-op
Proportion of subjects that require electrocautery or any other intervention post catheter removal. | 7 days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra Sabnis, MD, Principal Investigator — Muljibhai Patel Urological Hospital
Locations (1):
- Muljibhai Patel Urological Hospital, Nadiād, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided